CLINICAL TRIAL: NCT02296359
Title: Vaccination Response in Individual Monozygotic Twins
Status: Terminated | Type: Observational
Why Stopped: Insufficient enrollment
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, George Mias, Assistant Professor, Michigan State University
Other Study IDs: 14-848FM
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Individuality; Asthma; Immune System and Related Disorders
MeSH Terms: conditions — Asthma | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — If the volunteers agree,tissue is stored for usage in future research without identifiers. This includes cells from blood and saliva and extracted DNA, RNA and protein. The cells may be used to grow a new cell line that may be maintained in the laboratory.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Asthma Discordant Monozygotic Twins: This is a group where one of the monozygotic twins has asthma and the other is non-asthmatic. Influenza Vaccination will be performed for both cohorts.
  Interventions: Biological: Influenza Vaccination
- Non-Asthma Concordant Monozygotic Twins: This is a group where both of the monozygotic twins are non-asthmatic. Influenza Vaccination will be performed for both cohorts.
  Interventions: Biological: Influenza Vaccination

INTERVENTIONS:
Biological: Influenza Vaccination — The individuals will be followed to observe their immune system activation, following their vaccination with the standard influenza vaccine approved for the year by the FDA.

SUMMARY:
Respiratory viruses are known to be risk factors for asthma (e.g respiratory syncytial viruses, RSVs, and Human Rhinoviruses, HRVs, may induce bronchiolitis, and wheezing illnesses respectively). The common flu is also known to be a risk factor and the Centers for Disease Control and Prevention (CDC) recommends that asthmatics receive the annual flu vaccine, as a high-risk group for related asthma exacerbations. The investigators will be evaluating the variation in individual responses over time after controlled immune activation following influenza vaccination of monozygotic twins, both discordant for asthma, and concordant non-asthmatic. The transition from initial healthy to immune-system activated physiological states post vaccination will provide unprecedented molecular (omics) data on the molecular dynamics of immune response to vaccination, and novel insight into the flu response. The investigators will infer novel networks and pathways and as well as the dynamics of genes and mechanisms involved in asthma, flu vaccination, and individual responses, and correlate them to evaluated personalized genetic risks in the same study. The investigators will be able to also contrast the vaccination response in asthmatic and non-asthmatic individuals, in a longitudinal approach which has never been performed before using multiple-omics that included an immunization response.

DETAILED DESCRIPTION:
Asthma pathogenesis and exacerbations have been associated to multiple risk factors, particularly respiratory viruses. In children respiratory syncytial viruses (RSVs) may induce bronchiolitis, and Human Rhinoviruses (HRVs) also may induce wheezing illnesses. RSVs and HRVs are age dependent risk factors for asthma, with the influenza virus also considered a prominent risk factor in adults. The Center for Disease Control recommends influenza vaccination in asthmatics annually. Both HRV and RSV infections were detected in a pilot integrative personal omics investigation, and provided a unique temporal expression signature in the non-asthmatic subject, with the involvement of a common set of antigen and defense response genes, as well as immune related pathways. These observed patterns in addition to the results of the vaccination study will be used as a guide, to find differences in healthy versus asthmatic patients' pathway activations which will provide insights into the genes and mechanisms involved in asthma pathogenesis and immune response to influenza vaccination. The twin paradigm will allow us to control for multiple confounding factors and focus on the individual genetic and possible epigenetic variation. The investigators will be able to infer novel networks and pathways and get into the genes and mechanisms involved in asthma, flu vaccination, and individual responses, while evaluating personalized genetic risks compared to medical history in the same study.

Our primary investigation involves integrative multi-omics monitoring of individual monozygotic twins, healthy or discordant for asthma, following their flu vaccination, over a period of two annual vaccination cycles. The investigators will be collecting blood samples from monozygotic twin volunteers, for multiple time-points post influenza vaccination. The measurements will be repeated the following year after a second vaccination. Genomic sequencing will be used to evaluate the volunteer's genomic risks based on variants with known disease association. Full transcriptome (via RNA-Sequencing), proteome and metabolome profiling (via mass spectrometry) will be performed per time-point, as well as cytokine profiling. This will allow the dynamic monitoring of thousands of molecular components and their responses to vaccination, capturing both the initial innate response reaction in addition to the adaptive response and return to baseline. The study involves following responses in blood and saliva components after influenza vaccination. Two annual vaccinations will be considered, one per year for 2 years, and at 8 time points samples will be collected.

This study involves a simple blood draw, saliva collection, standard FDA-approved influenza vaccine administration and Spirometry.

ELIGIBILITY:
Inclusion Criteria:

Volunteers are eligible to participate in this study if both they and their twin sibling have agreed to participate. If after their enrollment in the study, one of the twin siblings decides to withdraw, then:

1. If one sibling withdraws during Year 1, the other sibling will be allowed to continue their participation in the study and to complete the current study Year. However they will not be included in the randomly selected applicants that will continue participation in Year 2 of the study.
2. If one sibling withdraws duringYear2, the other sibling will be able to conclude Year2 study activities. -

Exclusion Criteria:

1. Volunteer is under18.
2. Presence of any medical conditions that the study investigators believe will affect participation in the study or its results.
3. Presence of a mental incapacity and/or cognitive impairment that would prevent a subject from adequately understanding, or cooperating with, the study protocol.
4. Volunteers with any severe allergies (life-threatening) or that have ever had a life-threatening allergic reaction after a dose of flu vaccine, or have a known severe allergy to any part of this vaccine, will be advised not to participate.
5. If a potential subject has ever had Guillain-Barré Syndrome (a severe paralyzing illness, also called GBS), they will be advised not to get the influenza vaccine and be excluded from this study.

   * For female participants If they are already enrolled and become pregnant during this study, the investigators will temporarily withdraw them from the study from the day they become pregnant. If they would like to stay in the study, the investigators may continue their participation after their delivery.
   * If participants are not feeling well on the scheduled day of vaccination the investigators will suggest that they postpone the vaccination until they feel better. If they agree, the vaccination will be re-scheduled for a later date.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Monozygotic Twins over 18 years of age with and without asthma, without gender or ethnicity restrictions.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Integrated Omics profile | all time points (8 per year for 2 years per subject)
  The study will construct RNA-expression, protein profiles and small molecule profiles on immune cells as these change over time prior to and following immune activation by the vaccine. The collective temporal patterns will be used to classify immune response

CONTACTS AND LOCATIONS:
Overall Officials: George Mias, PhD, Principal Investigator — Michigan State University
Locations (1):
- Clinical and Translational Science Institute, East Lansing, Michigan, United States